CLINICAL TRIAL: NCT04163783
Title: A Phase 1 Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-BGB-3111 Following Single Oral Dose Administration in Healthy Male Subjects
Brief Title: Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-BGB-3111 in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BGB-3111-105
Record Dates: First submitted 2019-11-05; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
Keywords: Phase 1; Pharmacokinetics; Safety
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): Subjects will be administered a single oral dose of 320 mg of [14C]-BGB-3111
  Interventions: Drug: [14C]-BGB-3111; Drug: BGB-3111

INTERVENTIONS:
Drug: [14C]-BGB-3111 — 20-mg capsule containing ~200 μCi of [14C]-BGB-3111,
Drug: BGB-3111 — Three 20-mg capsules of BGB-3111 and three 80-mg capsules of BGB-3111

SUMMARY:
Phase 1 study in healthy subjects to determine the effect of an 8-hour fast from food on the pharmacokinetics of [14C]-BGB-3111.

DETAILED DESCRIPTION:
This study will be an open-label, non-randomized study to evaluate the pharmacokinetics of [14C]-BGB-3111 when administered in healthy male subjects following at least an 8-hour fast from food (not including water).

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18 and 65 years of age, inclusive, at Screening
2. Body mass index between 18.0 and 35.0 kg/m2, inclusive, at Screening
3. In good health, determined by no clinically significant findings from medical history,12-lead ECGs, or vital signs measurements
4. Clinical laboratory evaluations

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, infectious, dermatological, hepatic, renal, hematological, pulmonary, metabolic, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator [or designee]) prior to Check-in
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee) prior to Check-in
3. History of stomach or intestinal surgery or resection that could alter absorption or excretion of orally administered drugs prior to Check-in except that appendectomy and hernia repair will be allowed if it was not associated with complications
4. Abnormal liver function tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter: Plasma concentration of [14C]-BGB-3111 as measured by area under concentration-time curve (AUC) | Up to 13 days
Pharmacokinetic Parameter: Maximum Plasma Concentration (Cmax) of [14C]-BGB-3111 | Up to 13 days
Pharmacokinetic Parameter: Time To Maximum Plasma Concentration (Tmax) of [14C]-BGB-3111 | Up to 13 days
Pharmacokinetic Parameter: apparent terminal elimination rate constant (λZ) of [14C]-BGB-3111 | Up to 13 days
Pharmacokinetic Parameter: Half-life Period of (T1/2) of [14C]-BGB-3111 | Up to 13 days
Pharmacokinetic Parameter: apparent systemic clearance (CL/F) of [14C]-BGB-3111 | Up to 13 days
Pharmacokinetic Parameter: apparent volume of distribution during the terminal phase (Vz/F) of [14C]-BGB-3111 | Up to 13 days
Blood and plasma concentrations of total radioactivity: Maximum Plasma Concentration (Cmax) of [14C]-BGB-3111 | Up to 13 days
Blood and plasma concentrations of total radioactivity: Time To Maximum Plasma Concentration (Tmax) of [14C]-BGB-3111 | Up to 13 days
Blood and plasma concentrations of total radioactivity of [14C]-BGB-3111 as measured by area under concentration-time curve (AUC) | Up to 13 days
Blood and plasma concentrations of total radioactivity: apparent terminal elimination rate constant (λZ) of [14C]-BGB-3111 | Up to 13 days
Blood and plasma concentrations of total radioactivity: Half-life Period of (T1/2) of [14C]-BGB-3111 | Up to 13 days
Blood and plasma concentrations of total radioactivity: apparent systemic clearance (CL/F) of [14C]-BGB-3111 | Up to 13 days
Blood and plasma concentrations of total radioactivity: apparent volume of distribution during the terminal phase (Vz/F) of [14C]-BGB-3111 | Up to 13 days
Urinary recovery of total radioactivity of [14C]-BGB-3111 as assessed by the amount excreted in urine per sampling interval (Aeu) | Up to 13 days
Urinary recovery of total radioactivity of [14C]-BGB-3111 as assessed by the cumulative amount excreted in urine per sampling interval (Cum Aeu) | Up to 13 days
Urinary recovery of total radioactivity of [14C]-BGB-3111 as assessed by the percentage of drug or radioactive dose excreted in urine per sampling interval (%Feu) | Up to 13 days
Urinary recovery of total radioactivity of [14C]-BGB-3111 as assessed by the cumulative percentage of drug or radioactive dose excreted in urine (Cum %Feu) | Up to 13 days
Urinary recovery of total radioactivity as assessed by the renal clearance (CLR; for BGB-3111 only) | Up to 13 days
Fecal recovery of total radioactivity as assessed by the amount of [14C]-BGB-3111 excreted in feces per sampling interval (Aef) | Up to 13 days
Fecal recovery of total radioactivity as assessed by the cumulative amount of [14C]-BGB-3111 excreted in feces per sampling interval (Cum Aef) | Up to 13 days
Fecal recovery of total radioactivity as assessed by the percentage of radioactive dose excreted in feces per sampling interval (%Fef) | Up to 13 days
Fecal recovery of total radioactivity as assessed by the cumulative percentage of radioactive dose excreted in feces per sampling interval (Cum %Fef) | Up to 13 days
Mass balance | Up to 13 days
  Urine and fecal collection for Mass Balance Evaluation
Routes of elimination of [14C]-BGB-3111 | Up to 13 days
  Urine and fecal collection for Metabolite Profiling/Characterization

SECONDARY OUTCOMES:
Characterize and identify metabolites of [14C]-BGB-3111 | Up to 13 days
  plasma, urine, and feces collection
plasma and urine concentrations of BGB-3111 | up to 13 days
  plasma and urine collection
Number of Participants experiencing Adverse events (AEs) | up to 13 days
Number of Participants experiencing abnormal clinical laboratory evaluations | up to 13 days

CONTACTS AND LOCATIONS:
Overall Officials: William Novotony, MD, Study Director — BeiGene
Locations (1):
- Covance Clinical Research Unit, Inc.,, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes